CLINICAL TRIAL: NCT03676907
Title: Assessment of Single and Double Layer Suturation of Lower Segment Uterine Incision by Ultrasonography After Cesarean Section
Brief Title: Assessment of Single and Double Layer Suturation of Lower Segment Uterine Incision by USG After C/S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Erhan Demirdag, Academic, Director, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 237
Record Dates: First submitted 2018-09-11; First posted 2018-09-19 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Uterine Scar
Keywords: cesarean scar defect; single suturation technique; double suturation technique; myometrial thickness; uterine scar

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single layer suturation technique (No Intervention): in this arm we use single layer suturation technique to suture uterine incision
- double layer suturation technique (Experimental): in this arm we use double layer suturation technique to suture uterine incision
  Interventions: Procedure: double layer suturation technique

INTERVENTIONS:
Procedure: double layer suturation technique — in our clinic uterine incision is sutured by single layer suturation technique routinely. in this arm, we will use double layer suturation technique which is also accepted as valid suturation technique in obstetrics and gynecology textbooks
  Arms: double layer suturation technique

SUMMARY:
After 6 months of cesarean delivery, the investigators will compare uterine incision scar defects of single and double layer suturation of uterine incision by transvaginal ultrasonography.

DETAILED DESCRIPTION:
In our clinic, cesarean operation is performed with blunt and sharp dissections in the abdomen followed by transverse incision of the lower segment to the uterus. After uterotomy, the incision will be closed with single or double layer suture. The single layer suture technique will be performed with suturing by taking approximately 1 cm of tissue from the upper and lower segments where the mucosa and muscular layer are stitched together and locking them continuously at intervals of about 1 cm. On the first layer of the double layer suture technique, about 0.5 cm of tissue is taken from the upper and lower segments and the mucosa is closed by locking about 1 cm intervals. On the second layer, about 1 cm of tissue is taken from lower and upper segments of the muscle layer and both sides will be sutured with continue non-locking suture technique. The uterotomy incision will be closed with multifilament, synthetic, braided, suture that absorbable in about 60-90 days. In both groups prophylactic intramuscular 1 gr Cefazolin and 20 intravenous units of oxytocin will be administered intravenously.

Randomization will be done according to the patient's ID numbers. Patients who have a single digit of the end of ID number will be closed with continuous locking with suture, and patients who have a single digit of the end of ID number will be closed with double suture. The suture technique used and the number of additional hemostatic sutures will be obtained from the operation note. In addition, demographic characteristics of the patients, duration of operation, hemoglobin changes within 24 hours post-operatively, infant birth weight, hospitalization time, estimated blood loss during surgery will be examined in the study. The estimated blood loss will be recorded from the level of the initial aspirator bag after the surgery.

Enrolled patients will be called for control 6 months after surgery. It will be evaluated by a single obstetrician in a supine position under standard conditions, with empty bladder, with transvaginal ultrasonographic device. Measurements will be made when the endometrium, lower uterine segment and cervix are visible in the sagittal section of the uterus during transvaginal ultrasonography. Scar defect will define as a hypoechoic wedge-shaped image that causes discontinuity in the structure of the endometrium which extending downward from the anterior line to the serosa. The width and depth of the sagittal plane of the defect and the axial length of the axial plane will be measured. Ultimately, these measurements will be taken volumetrically.

ELIGIBILITY:
Inclusion Criteria:

* Those who are agreeing to participate in the study
* Planned or elective caesarean section
* The term singular pregnancies between 37 weeks 0/7 days - 41weeks 6/7 days of gestation that will be delivered on cesarean section without emergency conditions will be included in the study.

Exclusion Criteria:

* Not accepting to participate in the work
* Emergency cesarean
* Multiple pregnancy
* Diabetic patients
* Past uterine surgery
* Uterine malformation
* The infectious process (local, uterine or systemic)
* If surgeon needs additional two more hemostatic suturation during cesarean section.
* Women with connective tissue disease will not be included in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 56 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Comparing defective volume of myometrium at the location of cesarean section scar in double layer suturation technique and single layer suturation technique | Over 6 months period after cesarean section
  The volume measurement will be obtained ultrasonographically as a result of the width and depth measured on the sagittal plane of the defect as described by the formula of π x 4/3 multiplied by the length which will be imaged on the axial section of the uterus. The length of myometrial tissue that extends perpendicularly from the lower end of the scar defect to the serosa, ie the distance between the inner and outer edges of the cesarean scar, will be assessed and measured as the residual myometrial thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Erhan DEMİRDAĞ, MD. Academic, Study Director — Ankara Gazi Üniversitesi Tıp Fakültesi Hastanesi; Anıl Doğukan Tutal, MD, Principal Investigator — Ankara Gazi Üniversitesi Tıp Fakültesi Hastanesi; Recep Onur Karabacak, MD. Academic, Study Chair — Ankara Gazi Üniversitesi Tıp Fakültesi Hastanesi
Locations (1):
- Gazi University Faculty of Medicine, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Raine-Fenning N, Jayaprakasan K, Clewes J, Joergner I, Bonaki SD, Chamberlain S, Devlin L, Priddle H, Johnson I. SonoAVC: a novel method of automatic volume calculation. Ultrasound Obstet Gynecol. 2008 Jun;31(6):691-6. doi: 10.1002/uog.5359. PMID 18484679